CLINICAL TRIAL: NCT00160186
Title: Double-Blind, Multicenter, Randomized, Placebo-Controlled, Parallel-Group Study to Investigate the Effect of Creon 25000 Minimicrospheres on Body Mass Index (BMI) in Patients After Gastrectomy
Brief Title: Gastrectomy Study: Study to Investigate the Effect of Creon 25000 Minimicrospheres on Body Mass Index (BMI) in Patients After Gastrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Gregor Eibes, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S245.4.007
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Gastrectomy
MeSH Terms: interventions — Pancreatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Pancreatin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pancreatin — 2 capsules Pancreatin with 25 000 lipase units per main meal (3 meals) and 1 capsule per snack (2-3 snacks)
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to investigate BMI and the nutritional parameters of Creon (pancreatin) versus placebo after a total or subtotal gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Males or females
* Age >= 18 years
* Total or subtotal gastrectomy
* Females having negative pregnancy test or being surgically sterile or 1 year postmenopausal; women of childbearing age must use effective birth control.

Exclusion Criteria:

* Diseases or conditions limiting the participation in, or completion of, the study
* Progressive tumors/metastasis
* Complications leading to insufficient peroral nutrition
* Known allergy to pancreatin
* Known exocrine insufficiency
* Experimental drug intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-12; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted body mass index (BMI) after 6 months therapy | 6 months

SECONDARY OUTCOMES:
Effect on body composition, on stool fat, on the coefficient of fat absorption, stool weight, quality of life (Qol), clinical symptoms (gastrointestinal), data from the diary, Elastase | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (9):
- Site 9, Odense, Denmark
- Site 10, Tampere, Finland
- Norway (3):
  - Site 1, Bergen
  - Site 2, Fredrikstad
  - Site 3, Tromsø
- Sweden (4):
  - Site 5, Linköping
  - Site 7, Malmo
  - Site 6, Stockholm
  - Site 8, Stockholm